CLINICAL TRIAL: NCT00438295
Title: Effect of Temperature Control During Dialysis Treatment With Glucose in Dialysis Water in Patients With Chronic Renal Failure
Brief Title: Temperature Control During Dialysis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED.RES.2007.03.EBP
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2007-09

CONDITIONS: Renal Failure, Chronic
Keywords: glucose in dialysis water, dialysis treatment, temperature
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: temperature control

SUMMARY:
The purpose is to measure the effect of glucose in the dialysis water on blood pressure, pulse rate, and plasma glucose with and without body temperature control

DETAILED DESCRIPTION:
To clarify the influence of temperature in dialysis water on blood pressure and vasoactive hormones

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years,
2. both men and women,
3. chronic renal failure and dialysis treatment for at least three months

Exclusion Criteria:

1. Heart failure,
2. Lung insufficiency,
3. Chronic liver disease,
4. Diabetes mellitus,
5. Malignant disease,
6. Nephrotic syndrome,
7. Lack of compliance,
8. Unwillingness til participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Effect of temperature control on blood pressure, pulse rate and blod glucose during dialysis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro
Locations (1):
- Holstebro Hospital, Holstebro, Denmark